CLINICAL TRIAL: NCT02618603
Title: The Effectiveness of Ultrasound Guided Sub-acromial Bursa Injection With Botulinum Toxin A in for Refractory Shoulder Pain After Stroke.
Brief Title: Botulinum Toxin A for Shoulder Pain After Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, TAO WU, MD, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016137443; 2016137443 (Other Grant/Funding Number: Medical Science and Technology projects of Zhejiang Provincial Health Department)
Record Dates: First submitted 2015-11-27; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Stroke; Pain
Keywords: Stroke; Should pain; Botulinum Toxin
MeSH Terms: conditions — Stroke; Pain | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BoNT-A treatment group (Experimental): Ultrasound guided sub-acromial bursa injection with BoNT-A (100 u);
  Interventions: Drug: Botulinum toxin A
- Triamcinolone acetonide treatment group (Active Comparator): Ultrasound guided sub-acromial bursa injection with Triamcinolone acetonide (40mg)+1% Lidocaine 2 ml;
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Botulinum toxin A
  Other Names: BoNT-A
  Arms: BoNT-A treatment group
Drug: Triamcinolone Acetonide
  Arms: Triamcinolone acetonide treatment group

SUMMARY:
Shoulder pain after stroke is a very common, causing significant morbidity disease. Subacromial and subdeltoid (SASD) bursitis are common causes of pain or disability of the shoulder joint in stroke patients. Traditional therapeutic approaches for the shoulder pain therapy including pharmacotherapy, injection therapy, physical therapy, and behavioural modification. Unfortunately, these therapy methods may not be effective in many patients and long term benefit after treatment is transient, the outcomes may also be incomplete or non-existent. Botulinum toxin A (BoNT-A) is a neurotoxin that can inhibit not only the acetylcholine at the neuromuscular junctions but also other neurotransmitters such as glutamate, substance P and calcitonin gene related peptide, all of which have been indicated in pain transmission. Despite the therapeutic benefit of BTX in alleviating painful muscle spasms, its efficacy in SASD bursitis conditions is less clear. So we perform this study to examine the efficacy of ultrasound guided SASD injection with BoNT-A in reducing refractory shoulder pain after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke patients with pain around the shoulder or lateral deltoid area and deteriorated during active or passive overhead activity;
2. Neer and/or Hawkins tests (+);
3. NRS>5 at rest;
4. Symptoms lasted for at least for 2 months and were unresponsive to analgesic medication or physical therapy for 1 month.
5. Subjects voluntarily sign the informed consent.
6. Age between 18 and 80 years old. -

Exclusion Criteria:

1. Received earlier subacromial injections of corticosteroids or botulinuim toxin in the last 6 months;
2. Shoulder fracture, glenohumeral osteoarthritis, bone tumors or osteonecrosis in plain radiographs.
3. Known allergy or sensitivity to study medication or its components.
4. Infection or dermatological condition at the injection sites.
5. Any medical condition that may put the subject at increased risk with exposure , including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might have interfered with neuromuscular function.
6. QTc criteria: QTc ≥ 450 millisecond (msec) or≥480msec for subjects with Bundle Branch Block-values based on either single electrocardiogram (ECG) values or triplicate ECG averaged QTc values obtained over a brief recording period
7. Liver function tests: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥2xULN; alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
8. Concurrent use of aminoglycoside antibiotics or other agents that might interfere with neuromuscular function.
9. Patients with severe cognitive impairment or neurological diseases affecting the implementation or evaluation of the test, and drug-dependent patients.
10. Presence of clinically unstable severe cardiovascular, renal or respiratory disease
11. Researchers believe there are other factors unfit to participate in this study of patients.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of pain score (Numeric Rating Scale, NRS) | The outcome will be undertaken at weeks 0 (baseline), 1,2,4,8, and 12 weeks after injection.

SECONDARY OUTCOMES:
Passive and/or active shoulder range of motion. | The outcome will be undertaken at weeks 0 (baseline), 1,2,4,8, and 12 weeks after injection.
Change from baseline of should muscle modified Ashworth scale assess (MAS) | The outcome will be undertaken at weeks 0 (baseline), 1,2,4,8, and 12 weeks after injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Lee JH, Lee SH, Song SH. Clinical effectiveness of botulinum toxin type B in the treatment of subacromial bursitis or shoulder impingement syndrome. Clin J Pain. 2011 Jul-Aug;27(6):523-8. doi: 10.1097/AJP.0b013e31820e1310. PMID 21368663
- [Result] McMahon HT, Foran P, Dolly JO, Verhage M, Wiegant VM, Nicholls DG. Tetanus toxin and botulinum toxins type A and B inhibit glutamate, gamma-aminobutyric acid, aspartate, and met-enkephalin release from synaptosomes. Clues to the locus of action. J Biol Chem. 1992 Oct 25;267(30):21338-43. PMID 1356988
- [Result] Bach-Rojecky L, Salkovic-Petrisic M, Lackovic Z. Botulinum toxin type A reduces pain supersensitivity in experimental diabetic neuropathy: bilateral effect after unilateral injection. Eur J Pharmacol. 2010 May 10;633(1-3):10-4. doi: 10.1016/j.ejphar.2010.01.020. Epub 2010 Feb 1. PMID 20123097
- [Result] Hsieh LF, Hsu WC, Lin YJ, Wu SH, Chang KC, Chang HL. Is ultrasound-guided injection more effective in chronic subacromial bursitis? Med Sci Sports Exerc. 2013 Dec;45(12):2205-13. doi: 10.1249/MSS.0b013e31829b183c. PMID 23698243
- [Result] Wu T, Song HX, Dong Y, Li JH. Ultrasound-guided versus blind subacromial-subdeltoid bursa injection in adults with shoulder pain: A systematic review and meta-analysis. Semin Arthritis Rheum. 2015 Dec;45(3):374-8. doi: 10.1016/j.semarthrit.2015.05.011. Epub 2015 May 21. PMID 26590864
- [Result] Wu T, Fu Y, Song HX, Ye Y, Dong Y, Li JH. Effectiveness of Botulinum Toxin for Shoulder Pain Treatment: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2015 Dec;96(12):2214-20. doi: 10.1016/j.apmr.2015.06.018. Epub 2015 Jul 17. PMID 26189200